CLINICAL TRIAL: NCT03618524
Title: Effect of Local Heat Stress Via Leg Bath on Artery Function
Acronym: HEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Maureen MacDonald, Professor; Dean, Faculty of Science, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HEAT
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Endothelial Dysfunction
Keywords: heat stress; endothelial function; hot water immersion; arterial stiffness
MeSH Terms: conditions — Heat Stress Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Lower limb hot water immersion
  Interventions: Other: Lower limb hot water immersion

INTERVENTIONS:
Other: Lower limb hot water immersion — Participants will undergo two interventions in separate visits: lower limb hot water (42 deg C) immersion up to the (1) ankles or (2) knees.

SUMMARY:
Arteries are flexible in their structure and function and change in response to a variety of factors. Endothelial cells, are the skin type cells that form a layer inside arteries, and they are very important for arterial health. When they work properly, they produce substances that make the artery enlarge and support a healthy environment; but when they do not work properly, they produce substances that make the artery constrict and lead to a harmful environment. We can measure the function of these cells using an ultrasound machine and a quick test. The application of heat has been shown to change the structure and function of arteries, but we need to understand how these changes happen before we can effectively use heat as a therapy. Limb heating protocols (e.g., leg bath), in contrast with whole-body heating modes (e.g., sauna), are appealing as therapies because they generally cost less and are easier to use; but evidence is needed to demonstrate that they work before widespread use can be considered. Imagine soaking your legs in a bathtub filled with warm water becoming part of the options you have for staying healthy. Clearly, there is a lot of potential for heat to be used as a therapy, particularly for people who are unable to, or have difficulty participating in other health interventions that are known to improve arterial, but we need to do this type of research before we are able to recommend warm foot baths for therapeutic purposes.

DETAILED DESCRIPTION:
A within-subjects interventional design will be used in a cohort of 16 young, healthy males and females between the ages of 18-35 years old. Interested individuals will be invited to the lab for a screening and familiarization visit, in which the brachial artery (BA) and superficial femoral artery (SFA) will be scanned to vet for ultrasound image quality and BA and SFA flow-mediated dilation tests will be performed to ensure participant tolerance during collection visits. According to current FMD guidelines, all qualified participants will be instructed to refrain from vigorous physical activity > 24 hours, alcohol and caffeine > 8 hours, and food > 6 hours prior to each of the two experimental visits. Participants will also be asked to ingest a wireless telemetry pill 2 hours prior to each of the two experimental visits. Upon arrival, basic anthropometric measures will be collected and hematocrit will be measured in duplicate with a finger prick blood sample equivalent to two 70 µl capillary tubes. Experimental visits will begin with 10 minutes of supine rest, while the participant is instrumented with skin temperature probes on the foot, calf, thigh, chest, and arm for measurement of skin temperature; single-lead ECG (Powerlab model ML795, ADInstruments, Colorado Springs, CO, USA) and non-invasive finger cuff (Finometer MIDI, Finapres, The Netherlands) for continuous heart rate and blood pressure monitoring. Following rest, BA and SFA FMD tests will be conducted to assess baseline endothelial function. Afterwards, single-point laser Doppler flowmetry focused on the forearm will be used to track skin blood flow continuously throughout heating. The heating protocol will involve participants immersing their lower limbs either up to the ankles or the knees in a 42 °C water bath for 45 minutes, in separate conditions. The order by which participants undergo these interventions will be randomized. Five minutes after the conclusion of the intervention, BA and SFA FMD tests will be conducted to assess endothelial function in the acute phase. BA and SFA blood velocities, blood flow turbulence, endothelial shear rate, and oscillatory shear index will be assessed before and during each of the interventions; and arterial stiffness defined as carotid-femoral pulse wave velocity (PWV) and common carotid artery (CCA) distensibility will be assessed before and after each of the interventions as additional outcomes. Participants will provide written informed consent prior to beginning any portion of the study.

ELIGIBILITY:
Inclusion Criteria:

Apparently health (i.e., no cardiovascular, musculoskeletal, or metabolic disease), 18-35 years old 18-35 years old Recreationally active (exercising 2-3 times per week)

Exclusion Criteria:

History of cardiovascular, musculoskeletal, or metabolic disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation | Up to 2 weeks
  Collected using vascular ultrasound and analyzed using semi-automated edge tracking software

SECONDARY OUTCOMES:
Endothelial shear stress | Up to 2 weeks
  Calculated using blood velocity and arterial diameter obtained from vascular ultrasound, and blood density and viscosity calculated using hematocrit
Pulse wave velocity | Up to 2 weeks
  Collected using applanation tonometry and analyzed using data acquisition software
Arterial distensibility | Up to 2 weeks
  Collected using ultrasound imaging and applanation tonometry, and analyzed using semi-automated edge tracking software and data acqusition software

CONTACTS AND LOCATIONS:
Overall Officials: Maureen J MacDonald, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University Vascular Dynamics Lab, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brunt VE, Howard MJ, Francisco MA, Ely BR, Minson CT. Passive heat therapy improves endothelial function, arterial stiffness and blood pressure in sedentary humans. J Physiol. 2016 Sep 15;594(18):5329-42. doi: 10.1113/JP272453. Epub 2016 Jun 30. PMID 27270841
- [Background] Brunt VE, Eymann TM, Francisco MA, Howard MJ, Minson CT. Passive heat therapy improves cutaneous microvascular function in sedentary humans via improved nitric oxide-dependent dilation. J Appl Physiol (1985). 2016 Sep 1;121(3):716-23. doi: 10.1152/japplphysiol.00424.2016. Epub 2016 Jul 14. PMID 27418688
- [Background] Carter HH, Spence AL, Atkinson CL, Pugh CJ, Naylor LH, Green DJ. Repeated core temperature elevation induces conduit artery adaptation in humans. Eur J Appl Physiol. 2014 Apr;114(4):859-65. doi: 10.1007/s00421-013-2817-2. Epub 2014 Jan 8. PMID 24399113
- [Background] Deanfield JE, Halcox JP, Rabelink TJ. Endothelial function and dysfunction: testing and clinical relevance. Circulation. 2007 Mar 13;115(10):1285-95. doi: 10.1161/CIRCULATIONAHA.106.652859. No abstract available. PMID 17353456
- [Background] Gimbrone MA Jr, Garcia-Cardena G. Endothelial Cell Dysfunction and the Pathobiology of Atherosclerosis. Circ Res. 2016 Feb 19;118(4):620-36. doi: 10.1161/CIRCRESAHA.115.306301. PMID 26892962
- [Background] Kellogg DL Jr. In vivo mechanisms of cutaneous vasodilation and vasoconstriction in humans during thermoregulatory challenges. J Appl Physiol (1985). 2006 May;100(5):1709-18. doi: 10.1152/japplphysiol.01071.2005. PMID 16614368
- [Background] Naylor LH, Carter H, FitzSimons MG, Cable NT, Thijssen DH, Green DJ. Repeated increases in blood flow, independent of exercise, enhance conduit artery vasodilator function in humans. Am J Physiol Heart Circ Physiol. 2011 Feb;300(2):H664-9. doi: 10.1152/ajpheart.00985.2010. Epub 2010 Dec 3. PMID 21131471
- [Background] Tinken TM, Thijssen DH, Hopkins N, Black MA, Dawson EA, Minson CT, Newcomer SC, Laughlin MH, Cable NT, Green DJ. Impact of shear rate modulation on vascular function in humans. Hypertension. 2009 Aug;54(2):278-85. doi: 10.1161/HYPERTENSIONAHA.109.134361. Epub 2009 Jun 22. PMID 19546374
- [Background] Wong BJ, Hollowed CG. Current concepts of active vasodilation in human skin. Temperature (Austin). 2016 Jun 21;4(1):41-59. doi: 10.1080/23328940.2016.1200203. eCollection 2017. PMID 28349094